CLINICAL TRIAL: NCT06290167
Title: A New 360° Dual-task Based Protocol for the Pre-clinical In-hospital and At-home Rehabilitation of Elderly: DUAL-Rehab
Acronym: DUAL-Rehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 30M201
Record Dates: First submitted 2023-10-06; First posted 2024-03-04 (Actual); Last update posted 2025-08-04 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 360° media (Experimental): All participants will be randomly assigned to 360° media or TAU condition
  Interventions: Device: 360° media
- Treatment As Usual (TAU) (Active Comparator): All participants will be randomly assigned to TAU or 360° media condition
  Interventions: Other: Treatment As Usual (TAU)
- In hospital sessions (Other): all participants will perform session in hospital
  Interventions: Other: In hospital sessions
- at home sessions (Other): all participants will perform session at home
  Interventions: Other: at home sessions
- Mild Cognitive Impairment (Other): half of the patients will have MCI
  Interventions: Other: Mild Cognitive Impairment
- Subjective Memory Complain (Other): half of the patients will have SMC
  Interventions: Other: Subjective Memory Complain

INTERVENTIONS:
Device: 360° media — sessions with head mounted display in hospital and sessions with tablet at home
  Arms: 360° media
Other: Treatment As Usual (TAU) — sessions of TAU rehabilitation in hospital and sessions TAU rehabilitation at home
  Arms: Treatment As Usual (TAU)
Other: In hospital sessions — sessions will be carried out under the supervision of a therapist
  Arms: In hospital sessions
Other: at home sessions — sessions will be carried out without the supervision of a therapist
  Arms: at home sessions
Other: Mild Cognitive Impairment — half of this group will perform the protocol with 360° videos and the other half will perform the TAU
  Arms: Mild Cognitive Impairment
Other: Subjective Memory Complain — half of this group will perform the protocol with 360° videos and the other half will perform the TAU
  Arms: Subjective Memory Complain

SUMMARY:
The main objective of this project is two-fold

1. to develop a Dual-Task training exploiting the potentiality of the 360° technology in terms of interactivity and ecological validity
2. to investigate its efficacy in improving the cognitive functioning in a randomized clinical trial for 2 different populations: subjects with subjective memory complaints and mild cognitive impairment.

Specifically, participants will follow an integrated training including 2 phases: 1)in-hospital rehabilitation, where subjects will be provided sessions of the training in immersive modality; 2)at-home rehabilitation, where older adults will be asked to perform at home the non-immersive version of the training using a tablet.

Expected outcome is an improvement in cognitive functioning (assessed with a complete neuropsychological battery) after the training, thus advancing literature about non-pharmacological interventions in the preclinical stages of dementia along with innovative technical instruments.

ELIGIBILITY:
Inclusion Criteria (group of SMC):

* > 65 years old
* self-reported memory complaints
* score on Mini-Mental State Examination greater than or equal to 27/30 (normal range)

Exclusion Criteria:

* no evidence of objective impairments on the neuropsychological testing, scores on the Clinical Dementia Rating < 0.5

Inclusion Criteria (group of MCI):

* > 65 years old
* a self-reported (or reported by a caregiver) cognitive decline
* an objective impairment on the neuropsychological testing
* scores on the Clinical Dementia Rating < 0.5.

Exclusion Criteria:

* no dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Cognitive functions | Immediately after the training experience
  Improvement in cognitive functioning assessed with a complete neuropsychological battery focused on different domains such as executive function, memory, and attention.
Motor functions | Immediately after the training experience
  Improvement in motor functioning assessed with specific test focused on balance, functional mobility, and walking speed

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, MI, Italy